CLINICAL TRIAL: NCT05966844
Title: Golden Age: Virtual Reality and Mindfulness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Idego srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Golden Age 01-2023
Record Dates: First submitted 2023-07-12; First posted 2023-08-01 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Psychological Wellbeing; Healthy Lifestyle
Keywords: healthy lifestyle; psychological wellbeing

STUDY DESIGN:
Intervention Model Description: The project will investigate the effects of a Mindfulness pathway in RV on factors that hinder the adoption of healthy eating behaviour in the elderly population. Six meetings of about 5-10 minutes each, one per week, are planned. A randomised controlled trial (RCT) is proposed with two groups:
  * An experimental group of 20 elderly people who will do the trial in the RV.
  * Another control group, again of the same size, which will simply fill out simply twice the same battery of tests: one at the beginning of the project and the other at the end.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness and Virtual Reality (Experimental): This group will receive questionnaires at the beginning and end of the trial. In addition, they will undergo six mindfulness sessions in virtual reality for about six weeks. One session per week of approximately 5-10 minutes.
  Interventions: Behavioral: Mindfluness and Virtual Reality
- No intervention (No Intervention): This group will only receive questionnaires at the beginning and end of the experiment

INTERVENTIONS:
Behavioral: Mindfluness and Virtual Reality — They will undergo six mindfulness sessions in virtual reality for about six weeks. One session per week of approximately 5-10 minutes.
  Arms: Mindfulness and Virtual Reality

SUMMARY:
The aim of the research is to identify innovative methodologies to improve the psychological well-being of ageing people.

DETAILED DESCRIPTION:
With regard to the objectives of the Golden Age project, a software of Immersive Virtual Reality (VR) for people over 65. The application aims to improve the psychological wellbeing of ageing people, facilitating the removal of barriers that may represent a risk factor with respect to the assumption of a healthy and correct nutrition.

In particular, the elderly will be exposed to naturalistic scenarios in Virtual Reality combined with Mindfulness audio tracks. The practice of Mindfulness in Virtual Reality will be used to prevent and intervene on depressive symptoms, stress and anxiety, which represent the main obstacles to the adoption of healthy behaviours in the elderly person.

ELIGIBILITY:
Inclusion Criteria:

* Average age over 64
* MMSE between 20 and 30
* Adequate vision and hearing to see scenarios and hear tracks
* sufficient ability to understand procedures and communicate with staff

Exclusion Criteria:

* High levels of depression combined with other psychological risk indices (such as suicidal thoughts)
* Current use of narcotics or substance abuse

Min Age: 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Change in levels of GAD-7 test scores | Two months
  The GAD-7 test is a validated test for the detection of generalized anxiety disorder. GAD-7 total score for the seven items ranges from 0 to 21. Higher scores mean worse outcome.
Change in levels of PHQ-9 test scores | Two months
  The PHQ-9 test is a validated test for the detection of depression. The PHQ-9 score ranges from 0 to 24. Higher scores mean worse outcome.
Change in Perceived Stress Scale test scores | Two months
  The Perceived Stress Scale (PSS) test is a validated test for detecting general stress levels. The minimum score is 0 and the maximum score is 40. Higher scores mean worse outcome.
Change in Mindful Awareness Attention Scale scores | Two months
  The Italian Adaptation of the Mindful Awareness Attention Scale is a questionnaire investigating the presence of mindfulness skills.The minimum score is 15 and the maximum score is 105. A high score indicates an improvement.

SECONDARY OUTCOMES:
Level of acceptance and usability of devices | Two months
  Through a specifically designed questionnaire, the extent to which the devices used are perceived as useful, easy to use and accepted will be assessed. Questions on a 5-point likert scale will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Di Natale, Principal Investigator — Idego srl
Locations (1):
- Idego srl, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
Clinical data obtained from psychological testing and socio-demographic data and any feedback collected during the trial will be shared.
Supporting Information: Study Protocol
Time Frame: Data will be available starting from October 2023 for five years.
Access Criteria: The data available on the research website (www.idego.it). A specific page will be create where researchers can download the raw data to perform any analysis.